CLINICAL TRIAL: NCT00868088
Title: A Clinical Trial of ALA Photodynamic Therapy for Treatment of Actinic Cheilitis in Patients With Squamous Cell Carcinoma of the Lip.
Brief Title: Photodynamic Therapy to Treat Actinic Damage in Patients With Squamous Cell Carcinoma (SCC) of the Lip
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Gary Rogers, MD, Tufts Medical Center Department of Dermatology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PDT for Lip
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Actinic Cheilitis; Squamous Cell Carcinoma In-situ (SCC-is); Squamous Cell Carcinoma (SCC); Photodynamic Therapy (PDT); Mohs Surgery
Keywords: AC; SCC; SCC-is; PDT; Mohs
MeSH Terms: conditions — Actinic cheilitis; Squamous Intraepithelial Lesions; Carcinoma, Squamous Cell

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALA + PDT (Active Comparator): Topical ALA will be applied to the entire lip surface and allowed to incubate for 60 minutes plus or minus 30 minutes. Blue light at a wavelength of 405-420 nm will be used for treatment at a dose of 1000 seconds.
  Interventions: Procedure: PDT prior to Mohs surgery
- placebo + PDT (Placebo Comparator): Topical placebo will be applied to the entire lip surface and allowed to incubate for 60 minutes plus or minus 30 minutes. Blue light at a wavelength of 405-420 nm will be used for treatment at a dose of 1000 seconds.
  Interventions: Procedure: PDT prior to Mohs surgery

INTERVENTIONS:
Procedure: PDT prior to Mohs surgery — Day 1: Screening and consent for this study. If eligible, a scouting biopsy will be obtained at 1 cm from the clinical border of the SCC for confirmation of AC.
  7-14 Days after consultation: PDT to all subjects in the study. If during treatment a subject requests to discontinue due to pain the treatment will be terminated.
  3-5 weeks after consultation: return for assessment. At this visit, the assigned treatment may be repeated if the treatment site is adequately healed. Re-treatment will only occur if there is persistent actinic damage.
  6-8 weeks after consultation: Mohs surgery will be performed as per routine. Following tumor removal a scouting biopsy will be taken at a site 1 cm from the wound site created by SCC removal. The current waiting time for non-urgent surgery is 8 weeks. Standard care is not being altered for subjects in the study, other then their receiving the PDT intervention.
  Photographs may be taken at each subject visit.

SUMMARY:
Our study is designed to evaluate the efficacy of photodynamic therapy (PDT) for treatment of actinic cheilitis (AC) and as an adjunct to Mohs surgery for squamous cell carcinoma (SCC) on the lips. This study will utilize an FDA approved PDT modality (DUSA, Inc., Wilmington, MA 01887) using topical 5-amino-levulinic acid (ALA) for photosensitization followed by exposure to a Blu-U light source emitting 405-420nm wavelength light.

DETAILED DESCRIPTION:
BACKGROUND:

SCC of the lip is commonly surrounded by extensive AC, which may affect part or all of the lip vermillion. While Mohs surgical technique with complete margin control is the preferred treatment for SCC at critical locations such as the lip, this technique is complicated by surrounding AC. AC and SCC in situ at the tumor edge make it difficult to achieve margins clear of dysplasia and as a result extra tissue beyond the invasive SCC often needs to be excised to ensure that the entire tumor is removed.

Non-surgical treatments when used alone to treat SCC give lower cure rates than surgical removal, and thus are not recommended as they place the subject at risk for recurrence and metastatic disease. Although one study reported high SCC clearance rates with PDT alone (24/25 SCCs histologically cleared), recurrence of 2 SCCs occurred and a metastasis to a LN was seen in one patient. (Kubler et al.)

Given that PDT has been shown to have significant efficacy for actinic keratoses and actinic cheilitis but is inadequate as primary treatment of lip SCC, we propose that PDT may be a useful adjunct to surgical resection, allowing for less extensive surgery after the dysplasia is addressed with PDT and potentially a lower recurrence rate. Although imiquimod and 5-FU are also used to treat cutaneous dysplasia, many favor PDT treatment due to its greater tolerability, shorter healing time, and more predictable host response.

There is significant data on the efficacy of PDT for treatment of actinic keratoses (AKs) and PDT is now FDA approved for treatment of AKs. (Piacquadio et al). Data on PDT for treatment of AC is much more limited, but small studies and case reports do indicate successful treatment of AC with regimens utilizing either topical 5-aminolevulinic acid (5-ALA), or a similar compound, methylaminopentanoate (MAL). The largest study with 5-ALA reports complete clinical clearance in 13/19 patients treated with 1 to 3 treatments of ALA plus Pulsed-dye laser (Alexiades). Sotiriou et al report that with two PDT treatments 8/10 patients had complete clinical and histologic clearance (Sotiriou). Case reports indicate similar success (Kodama; Stender). Efficacy has also been shown with MAL PDT. One study found that with two sessions of MAL + red light PDT complete histologic/ clinical clearance was seen in 7/15 cases of AC and partial clearance was seen in an additional 7/15 (Berking et al). Smaller studies and case reports have shown even higher response rates without clinical recurrence during short-term follow-up (Rossi et al; Hauschild et al). We have chosen 5-ALA plus blue light for PDT treatment in this study because it is FDA approved for treatment of AKs and ALA is available in the United States.

Specific Aims:

1. To determine whether pre-operative treatment of the lips with ALA PDT can reduce the size of post-surgical defects (scars) in subjects with AC and lip SCC
2. To determine whether ALA PDT applied to the lips can effectively clear actinic cheilitis (AC) and SCC in-situ (SCC-is) of the lip.
3. To assess the tolerability of ALA PDT for treatment of AC and SCC-is of the lips

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven squamous cell carcinoma of the lip
* Greater than 50% of lip affected by actinic cheilitis by physical exam at time of initial evaluation.
* Patients > 18 years of age
* Patients must be able to provide informed consent

Exclusion Criteria:

* Patients with history of photosensitivity
* Patients with medical conditions associated with photosensitivity, such as cutaneous porphyria or a collagen vascular disease
* Patients taking medications known to cause photosensitivity (tetracyclines, sulfonamides, phenothiazines, sulfonylurea hypoglycemic agents, thiazide diuretics, griseofulvin, and fluoroquinolones)
* Patients with hypersensitivity to porphyrins.
* Women who are pregnant or nursing
* No exclusion based on gender or race
* Patients who have received anti-neoplastic treatment such as imiquimod or 5-FU to the lips within 30 days of enrolling in this study.
* Patients simultaneously participating in another research study for management of SCC or actinic cheilitis
* Subjects that plan to use other forms of AC treatment prior to Mohs.
* Subjects that have an SCC requiring urgent (and sooner) Mohs surgery, including those tumors that are large (> 2cm or at the discretion of the Principle Investigator) and those subjects that are pregnant or have palpable lymph nodes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine whether pre-operative treatment of the lips with ALA PDT can reduce the size of post-surgical defects (scars) in patients with AC and lip SCC. | at time of Mohs

SECONDARY OUTCOMES:
To determine whether ALA PDT applied to the lips can effectively clear actinic cheilitis (AC) and SCC in-situ (SCC-is) of the lip. | at time of Mohs.
To assess the tolerability of ALA PDT for treatment of AC and SCC-is of the lips | at time of PDT and Mohs

CONTACTS AND LOCATIONS:
Overall Officials: Gary Rogers, M.D., Principal Investigator — Tufts Medical Center, Department of Dermatology
Locations (1):
- Tufts Medical Center, Department of Dermatology, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kubler AC, de Carpentier J, Hopper C, Leonard AG, Putnam G. Treatment of squamous cell carcinoma of the lip using Foscan-mediated photodynamic therapy. Int J Oral Maxillofac Surg. 2001 Dec;30(6):504-9. doi: 10.1054/ijom.2001.0160. PMID 11829232
- [Background] Piacquadio DJ, Chen DM, Farber HF, Fowler JF Jr, Glazer SD, Goodman JJ, Hruza LL, Jeffes EW, Ling MR, Phillips TJ, Rallis TM, Scher RK, Taylor CR, Weinstein GD. Photodynamic therapy with aminolevulinic acid topical solution and visible blue light in the treatment of multiple actinic keratoses of the face and scalp: investigator-blinded, phase 3, multicenter trials. Arch Dermatol. 2004 Jan;140(1):41-6. doi: 10.1001/archderm.140.1.41. PMID 14732659
- [Background] Alexiades-Armenakas MR, Geronemus RG. Laser-mediated photodynamic therapy of actinic cheilitis. J Drugs Dermatol. 2004 Sep-Oct;3(5):548-51. PMID 15552607
- [Background] Sotiriou E, Apalla Z, Koussidou-Erremonti T, Ioannides D. Actinic cheilitis treated with one cycle of 5-aminolaevulinic acid-based photodynamic therapy: report of 10 cases. Br J Dermatol. 2008 Jul;159(1):261-2. doi: 10.1111/j.1365-2133.2008.08607.x. Epub 2008 Jul 1. No abstract available. PMID 18489592
- [Background] Stender IM, Wulf HC. Photodynamic therapy with 5-aminolevulinic acid in the treatment of actinic cheilitis. Br J Dermatol. 1996 Sep;135(3):454-6. PMID 8949443
- [Background] Kodama M, Watanabe D, Akita Y, Tamada Y, Matsumoto Y. Photodynamic therapy for the treatment of actinic cheilitis. Photodermatol Photoimmunol Photomed. 2007 Oct;23(5):209-10. doi: 10.1111/j.1600-0781.2007.00299.x. PMID 17803601
- [Background] Berking C, Herzinger T, Flaig MJ, Brenner M, Borelli C, Degitz K. The efficacy of photodynamic therapy in actinic cheilitis of the lower lip: a prospective study of 15 patients. Dermatol Surg. 2007 Jul;33(7):825-30. doi: 10.1111/j.1524-4725.2007.33176.x. PMID 17598848